CLINICAL TRIAL: NCT01440530
Title: Technology Intervention for Diabetes Engagement & Self-Care (TIDES):Comparative Effectiveness Randomized Clinical Trial in Primary Care for Type 2 Diabetes to Improve Engagement, Knowledge, and Self-Care
Brief Title: Technology Intervention for Diabetes Engagement & Self-Care (TIDES)
Acronym: TIDES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Dlife (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010-0173
Record Dates: First submitted 2011-09-20; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Internet Education; Diabetes Education; Diabetes Self-Care; Diabetes Self-Management; Diabetes Behavior Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention (Experimental)
  Interventions: Behavioral: Educational Intervention
- Control Group (usual care) (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Educational Intervention — Following randomization to TIDES (N=117) or usual care (N=49), TIDES group was oriented to the multimedia online intervention including a dosed sequence of learning via email, video, slideshows, food solutions, expert questions and answers, and quizzes.
  Arms: Educational Intervention
Other: Usual Care — Following randomization to TIDES (N=117) or usual care (N=49), TIDES group was oriented to the multimedia online intervention including a dosed sequence of learning via email, video, slideshows, food solutions, expert questions and answers, and quizzes.
  Arms: Control Group (usual care)

SUMMARY:
The purpose of this 3 site, 24-week, Comparative Effectiveness Randomized Clinical Trial in Primary Care is to compare usual care to an online, multi-media, digital intervention for Persons with Type 2 Diabetes to Improve Engagement, Knowledge, and Self-Care.

DETAILED DESCRIPTION:
Objective: Technology shows promise to enhance standard care of diabetes with cost-effective, online lifestyle interventions. Compared to Primary Care (PC) Diabetes System of Care (control), the investigators hypothesized Technology Intervention for Diabetes Engagement & Self-Care (TIDES) would significantly improve diabetes knowledge and self-care.

Methods: Following Institutional Review Board (IRB) approval, physician letters were sent to patients with type 2 diabetes, age >18 years with HgA1c >8% identified via Electronic Health Record (EHR) of an integrated US health system to invite participation in a 3-site, 24-week diabetes study. Of the 270 with >1 week email/web use invited to the shared medical visit (SMV) orientation, 166 subjects provided written informed consent. Diabetes knowledge and self-care assessments, vital signs, HgA1c, fasting glucose and lipids were collected at baseline, 3 and 6 months. Following randomization to TIDES (N=117) or usual care (N=49), TIDES group was oriented to the multimedia online intervention including a dosed sequence of learning via email, video, slide shows, food solutions, expert questions and answers,and quizzes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus Type 2
* Geisinger Primary Care Provider
* Access to a computer

Exclusion Criteria:

* Severe medical problems that limits travel to primary care
* Diabetes Type 1
* Cognitive Impairment
* Taking anti-psychotic meds

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Diabetes Knowledge | 6 months
  Change from Baseline Total Score on Diabetes Knowledge Questionnaire(DKQ)at 6 months.The DKQ is the shortened 24-item version of the Diabetes Knowledge Questionnaire was derived from an original 60-item instrument to reduce participant burden.Scores on the 60-item and 24-item versions are well correlated (r=0.85).Collins,G.S.,et al.,Modification and validation of the Revised Diabetes Knowledge Scale. Diabet Med, 2011. 28(3):p.306-10. Fitzgerald,J.T.,et al.,The reliability and validity of a brief diabetes knowledge test.Diabetes Care,1998.21(5):p.706-10.

SECONDARY OUTCOMES:
Diabetes Self Care | 6 months
  Change from Baseline on Partners in Health Scale(PIH)at 6 months.PIH is a validated instrument to measure self-management. The 11 items cover capacity and motivation for behavior change scored on a 9-point scale,with zero as best response and 8 worst.Four factors explain ~80% of variance in PIH scores: knowledge,symptom management,coping and adherence.Petkov, J.,P. Harvey,and M. Battersby, The internal consistency and construct validity of the partners in health scale:validation of a patient rated chronic condition self-management measure. Qual Life Res, 2010. 19(7):p.1079-85.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret R Rukstalis, MD, Principal Investigator — Geisinger Clinic
Locations (3):
- United States (3):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Clinic - Gray's Woods, Port Matilda, Pennsylvania
  - Geisinger Clinic - Kistler, Wilkes-Barre, Pennsylvania

REFERENCES:
- See also: Geisinger Health System — http://www.geisinger.org